CLINICAL TRIAL: NCT07083921
Title: Effect of Dominant and Non-dominant Hand Load Carry on Dynamic Plantar Pressure
Brief Title: Effect of Load Carry on Dynamic Plantar Pressure
Acronym: handload
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medipol University (Other)
Responsible Party: Principal Investigator, Hande YAZICI, Lecturer, Medipol University
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Screening
Other Study IDs: HIsci
Record Dates: First submitted 2025-06-13; First posted 2025-07-24 (Actual); Last update posted 2025-07-24 (Actual); Status verified 2025-06

CONDITIONS: Plantar Pressure Distrubution
Keywords: Dominant Hand; Non-Dominant Hand; load; dynamic plantar pressure
MeSH Terms: interventions — Gait Analysis

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Dominant hand (Experimental): Participants are evaluated only once.
  Interventions: Device: plantar pressure

INTERVENTIONS:
Device: plantar pressure — Healthy individuals carry loads with their dominant and non-dominant hands.
  Other Names: gait analysis

SUMMARY:
The aim of the study was to investigate the effect of loads carried with the dominant and non-dominant hand on dynamic plantar pressure parameters in healthy individuals.Participants were required to be between the ages of 20 and 55 years, and to be free from systemic, neurological, orthopaedic or chronic diseases. Individuals with physical or mental disabilities, balance problems, a risk of falling, knee or wrist-hand joint instability, or who were pregnant, were excluded from the study.

H1:Carrying load on the dominant hand increases dynamic plantar pressure parameter values.

H0: Carrying load in the dominant hand does not change the dynamic plantar pressure parameter values.

DETAILED DESCRIPTION:
Background: Individuals carry loads with their right or left hand due to their daily life activities. The load carried causes biomechanical differences on the body.

Research Question: The aim of the study was to investigate the effect of loads carried with the dominant and non-dominant hand on dynamic plantar pressure parameters in healthy individuals.

Method: 20 healthy participants aged 20-55 years participated in the study voluntarily. The participants were asked to walk at least six laps at normal walking speed while carrying a load weighing 4 kg with their right and then their left hands. The Sensor Medica pedobarography device was used to evaluate dynamic plantar pressure.

ELIGIBILITY:
Inclusion Criteria:

* between the ages of 20-55
* without any systemic, neurological, orthopaedic and chronic diseases

Exclusion Criteria:

* pregnant,
* physical and mental problems
* having balance problems and high risk of falling
* with joint instability

Ages: 20 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Actual)
Dates: Start 2021-01-15 (Actual); Primary Completion 2021-10-15 (Actual); Study Completion 2021-10-15 (Actual)

PRIMARY OUTCOMES:
Plantar Pressure | Baseline
  Plantar pressure will be measured with a baropodometer. The maximum pressure occurring at the time of measurement during load bearing shall be evaluated.

CONTACTS AND LOCATIONS:
Locations (2):
- Turkey (Türkiye) (2):
  - Istanbul Medipol University, Beykoz, Istanbul
  - Istanbul Medipol University, Istanbul, Istanbul

IPD SHARING:
Plan to Share IPD: No